CLINICAL TRIAL: NCT01458925
Title: Feasibility, Multi-center Prospective Study of Check-Cap's P1 Capsule System in Patients Eligible for ColoRectal Cancer [CRC] Screening
Brief Title: Feasibility of Check-Cap's P1 Capsule System Screening
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: All trials ojectives were met
Sponsor: Check-Cap Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CL-SY-01-0091
Record Dates: First submitted 2011-10-21; First posted 2011-10-25 (Estimated); Last update posted 2019-02-04 (Actual); Status verified 2019-01

CONDITIONS: ColoRectal Cancer; Colonic Polyps
Keywords: Colorectal cancer; Colonic polyps
MeSH Terms: conditions — Colorectal Neoplasms; Colonic Polyps

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- P1 capsule and screening Cscopy (Other): Male and female patients older than 40 and younger than 75 years old who volunteer for the experiment and qualify with the inclusion / Exclusion criteria.
  The P1 Check-Cap capsule will be ingested by all participants. After the Capsule test, they will be referred for optical colonoscopy as part of the study
  Interventions: Device: The P1 Check-Cap capsule

INTERVENTIONS:
Device: The P1 Check-Cap capsule — The P1 Check-Cap capsule will be ingested by all participants. After the Capsule test, they will be referred for optical colonoscopy as part of the study

SUMMARY:
Prospective, Single arm, Multi-Center

1. To establish the safety and preliminary efficacy of the Check-Cap System in patients with negative FOBT (Fecal Occult Blood Test)
2. To collect data about the overall imaging of the colon internal surface during the passage of the capsule
3. To develop a correlation map between the imaging of the polyps by optical colonoscopy vs. the images of same polyps by the Check-Cap capsule vs. the imaging of same polyps by CT Colonography [CTC] (in patients which were referred after positive CTC examination)

DETAILED DESCRIPTION:
Study Title:

Outside USA [OUS] Pilot Multi-center prospective feasibility study

Objectives:

Primary:

To establish the safety and preliminary efficacy of the Check-Cap System in patients with negative FOBT (Fecal Occult Blood Test) or FIT

Secondary:

* To evaluate the safety of the device in terms of total and segmental transit time and to study the effect of the presence of polyps and variable colon dimensions on these parameters.
* To monitor the functionality of the activation mechanism and of the scanning circuitry (transmitter detectors).
* To collect data about the overall imaging of the colon internal surface during the passage of the capsule
* To develop a correlation map between the imaging of the polyps by optical colonoscopy vs. the images of same polyps by the Check-Cap capsule vs. the imaging of same polyps by CT Colonography (in patients which were referred after positive CTC examination)
* To estimate the total radiation exposure to each patient.
* To measure the distribution of the contrast material within the colon.

Design:

Prospective, Single arm, Multi-Center

Patient population:

Group A - First in Man:

Male and female subjects older than 40 and younger than 75 years old that are eligible for CRC screening and meet the eligibility criteria for study enrollment.

The study population will be enriched with up to 45 patients with known polyps detected by CTC or colonoscopy, in addition to 15 patient of the device's normal cohort.

All patients that are eligible for enrollment in the study will be tested by FOBT (Fecal Occult Blood Test) After the Capsule test, they will be referred for optical colonoscopy as part of the study

Group B - CE Pilot:

Male and female subjects older than 45 and younger than 75 years old that are eligible for CRC screening and meet the eligibility criteria for study enrollment.

All patients that are eligible for enrollment in the study will be tested by FIT ,. After the Capsule test they will be referred for optical colonoscopy Consenting patients with negative FIT testing scheduled for clinically-indicated optical colonoscopy without contraindication to either Check-Cap System imaging or optical colonoscopy, and able to undergo the bowel preparation necessary for optical colonoscopy.

Sample Size:

Total of 100 patients in both groups: A:3-5 + B: 55-57 subjects.

Study Procedure:

1. st visit - recruitment and screening meeting with the Principal Investigator [PI]. Subject will receive the FIT test kit with detailed instructions for executing the test.
2. nd visit - The FIT kits will be analyzed in order to diagnose the presence of blood in the stool.

   If the bowel log form is complete and the bowel frequency is not less than once per 2 days the subject will be asked to sign the Informed Consent Form [ICF] for ingesting the capsule.
3. rd visit - Subject will ingest the capsule and continue ingestion of contrast material.
4. th visit - Subjects will return to the PI with the excreted capsule which is expected within 24-100 hours after ingestion.
5. th visit - All patients will undergo standard bowel preparation and optical colonoscopy between 10 and 30 days following imaging with the Check-Cap System.

ELIGIBILITY:
Inclusion Criteria:

* Male or female between 40 and 75 years of age.
* Subject is generally in good health.
* Subject is ready to undergo FOBT or FIT and Colonoscopy.
* Subject agrees to sign the informed consent.

Exclusion Criteria:

* Subject has any known Gastro Intestinal [GI] related symptoms, complaints or GI diseases.
* Subject is contraindicated from performing colon cleansing (bowel prep.)
* Subject has cancer or other life threatening diseases or conditions.
* Female subject is pregnant.
* Subject underwent any abdominal surgery.
* Morbid Obese (BMI > 40) subject.
* Subject has known drug abuse or alcoholism problem.
* Subject is under custodial care.
* Subject is currently or will be participating in other clinical study within 30 days prior to Check-Cap procedure

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 143 (Actual)
Dates: Start 2011-11-20 (Actual); Primary Completion 2018-09-16 (Actual); Study Completion 2019-01-02 (Actual)

PRIMARY OUTCOMES:
safety - transit time (less than 300 hours) | after each subject (once the capsule in excreted, typically 30-80 hours)
  To evaluate the safety of the device in terms of total and segmental transit time and to study the effect of the presence of polyps and variable colon dimensions on these parameters. The measured effect is the correlation of the capsule transit time (hours) with the number of polyps and their size (in mm).

SECONDARY OUTCOMES:
Colon Capsule correlation map (Empirical, qualitative) | end of study (anticipted within 12 months)
  To develop a correlation map between the imaging of the polyps by optical colonoscopy vs. the images of same polyps by the Check-Cap capsule vs. the imaging of same polyps by CT Colonography (in patients which were referred after positive CTC examination). No quantitative data here, only qualitative comparison between the scanning of the inner surface of the colon by the 3 independedt imaging modalities. No statistical plan or sample size justification would be provided, as is convention for pilot studies.

CONTACTS AND LOCATIONS:
Overall Officials: Yoav Kimchy, Ph.D.,, Study Chair — yoav.kimchy@check-cap.com
Locations (1):
- Tel Aviv Sorasky Medical Center, Tel Aviv, Israel

IPD SHARING:
Plan to Share IPD: No